CLINICAL TRIAL: NCT06259838
Title: Oral Cavity Squamous Cell Carcinoma and Readmission: Rates, Causes, and Risk Factors.
Status: Completed | Type: Observational
Sponsor: Abdulsalam Alqutub (Other)
Responsible Party: Sponsor-Investigator, Abdulsalam Alqutub, Dr, King Abdulaziz University
Organization: King Abdulaziz University (Other)
Other Study IDs: KingAbdulazizUn
Record Dates: First submitted 2024-02-07; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Oral Cavity Squamous Cell Carcinoma; Readmission
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
We sought to comprehend the rates and causes of unplanned hospital readmission within 60 days following oral cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* all patient underwent oral cancer surgery in king Abdulaziz University hospital

Exclusion Criteria:

* significant missing data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patient underwent oral cancer surgery in king Abdulaziz University hospital
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
rate of readmission | 60 days after discharge
  the number of readmitted patients within 60 days following oral cancer surgery

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No